CLINICAL TRIAL: NCT04109703
Title: High Level Pulsed Heat Versus Low Level Steady Heat in Subjects With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soovu Labs Inc. (Industry)
Collaborators: Northern California Research Corporation (Other); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201969K
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Results first posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-11

CONDITIONS: Chronic Pain; Low Back Pain; Heat; Analgesia
Keywords: chronic pain; low back pain; heat; thermal; analgesia
MeSH Terms: conditions — Chronic Pain; Low Back Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: Double blinded, randomized, active placebo controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded with a control condition using a low level heating (37 degree C) device. The active experimental device used heast that intermittently pulsed to 45 degrees C.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High level pulsed heat (Active Comparator): Subjects randomized to this arm received a generation 5 device (Soovu Labs Inc.) that produced 30 minutes of heat. The heat was delivered as waves peaking at 45° C.
  Interventions: Device: High Level Pulsed Heat delivered by Generation 5 devices from Soovu Labs Inc.
- Low level steady heat (Placebo Comparator): Subjects randomized to this arm received an identical generation 5 device (Soovu Labs Inc.) that produced 30 minutes of heat. The heat was delivered in a steady manner at 37° C.
  Interventions: Device: Low Level (37 degrees C) delivered by the control device Generation 5 devices from Soovu Labs Inc.

INTERVENTIONS:
Device: High Level Pulsed Heat delivered by Generation 5 devices from Soovu Labs Inc. — The Soovu Labss Inc. battery powered device is a one inch diameter heating pod that attaches to the user via a ring system. The device may be programmed to deliver a wide variety of treatment algorithms. Control of the devices are through a phone-based bluetooth connection. For this study the treatment algorithm used for subjects in this arm (experimental) used a temperature that was ramped from skin temperature to a peak temperature of 45° C and cycled for 30 minutes.
  Other Names: Experimental arm
  Arms: High level pulsed heat
Device: Low Level (37 degrees C) delivered by the control device Generation 5 devices from Soovu Labs Inc. — The Soovu Labs Inc. battery powered device is a one inch diameter heating pod that attaches to the user via a ring system. The device may be programmed to deliver a wide variety of treatment algorithms. Control of the devices are via a phone-based bluetooth connection. For this control arm of the study the treatment algorithm held a steady temperature of 37 degrees C for a 30 minute period.
  Other Names: Control arm
  Arms: Low level steady heat

SUMMARY:
This study is a double blinded randomized active placebo controlled trial in subjects with chronic low back pain. The trial compares pain relief by a device that delivered high level pulsed heat (45 °C) to pain relief delivered by a steady heat lower temperature device (37 °C). The hypothesis is that the high temperature pulsed heat device will produce significantly better pain relief as compared to the lower level steady heat device. The secondary hypothesis is that pain relief will occur faster in the high pulsed heat device as compared to the control device.

DETAILED DESCRIPTION:
1. This study will be conducted under Good Clinical Practice (GCP) guidelines and suitable for FDA submission in order to obtain claims such as, "provides temporary pain relief for people with chronic lower back pain."
2. The study is designed as a randomized double blinded two arm placebo controlled trial.
3. The active arm (N=50) receives two active Series 5 heating units (Soovu Labs Inc.) that pulse heat to 45ºC (113ºF). The active Series 5 placebo arm (N=50) gets two identical appearing units (Soovu Labs Inc.) that produce low level of heat at 37ºC (96.8 ºF). For reference skin temperature is about 33 ºC and room temperature 23 ºC.
4. The study hypothesis is that in subjects with chronic low back pain, the active heating device group will show a statistical improvement in pain scores as compared to the active placebo group as measured by the primary outcome measure, the Numeric Pain Scale (NPS).
5. Subjects will be told the study is examining the pain relieving effectiveness of two different levels of heat.
6. Subjects must have chronic low back pain with a pretreatment level of pain 4 or greater on a 0-10 point scale. By definition chronic low back pain is a condition that has been present for at least 6 months and must be present more days than not over the course of a week.
7. No use of pain medications during the four hour trial. However, pain medications including schedule IIIs can be taken up to 30 minutes before the start of the trial. Medications permitted during the trial include medications such as tramadol, codeine, NSIADs, gabapentin and acetaminophen. Non-pain medications for medical indications are permitted at any time. Subjects taking schedule II opioids are excluded from the study. Schedule II opioids include oxycodone, hydromorphone, hydrocodone, fentanyl and methadone.
8. Ages 22 through 70 inclusive.
9. Exclusion criteria- sciatica if present must be rated significantly less than the non -radiating component of the low back pain, pregnancy, skin lesions such as open skin or sores, scar tissue, skins grafts, old burns over the treatment area or neuropathic sensory loss over the treatment site.
10. Pre-treatment assessments include, Numeric Pain Scale, and a pre-study questionnaire (history, treatment preferences, short form Brief Pain Inventory, and short form Magill).
11. Each treatment session lasts approximately 30 minutes with pain assessments throughout using NPS (primary outcome measure). Secondary outcome measures include measures of comfort and willingness to endorse their treatment.
12. All subjects are followed for a 4 hour post treatment period with intermittent pain assessments (NPS).
13. At the end of the post treatment period, subjects complete a post study usability questionnaire and a blinding questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic low back pain. By definition chronic low back pain is a condition that has been present for at least 6 months on more days than not. If there is a radiating component of the low back pain the radiating component must have a pain rating less than the non-radiating component of the low back pain.
2. Subjects must have pretreatment level of pain 4 or greater.
3. Ages 22 through 70 inclusive
4. Non pain medications are permitted as needed for conditions such as hypertension, diabetes, heart disease etc.
5. Medications such as tramadol, codeine, NSIADs, gabapentin and acetaminophen are not permitted during the trial but may be included under the discretion of the study physician.
6. Subjects must have a reliable method for clinic contact and follow-up.

   -

Exclusion Criteria:

1. Sciatica or radicular pain without non-radiating low back pain, cancer, radicular pain greater than the non-radiating component of low back pain, pregnancy, skin lesions such as open skin or sores, scar tissue, skins grafts, old burns over the treatment area.
2. Medications including oxycodone, hydromorphone, hydrocodone, fentanyl and methadone are excluded from the trial but may be included under the discretion of the study physician. Such decisions will be documented should they occur.

   -

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — any gender eligible
Enrollment: 100 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: charles chabal, MD, Principal Investigator — Soovu Labs Inc.
Locations (1):
- Northern California Research Institute, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- High Level Pulsed Heat: Subjects randomized to this arm received a generation 5 device (Soovu Labs Inc.) that produced 30 minutes of heat. The heat was delivered as waves peaking at 45° C.
  Generation 5 device Soovu Labs Inc.: The Soovu Labs Inc. battery powered device is a one inch diameter heating pod that attaches to the user via a ring system. The device may be programmed to deliver a wide variety of treatment algorithms. Control of the devices are through a phone-based bluetooth connection. The treatment algorithm used for all subjects in this arm pulsed heat to a temperature of 45 degrees C.
- Low Level Steady Heat: Subjects randomized to this arm received an identical device (Soovu Labs Inc.) that produced 30 minutes ot heat. The heat was delivered in a steady manner at 37° C.
  Generation 5 device Soovu Labs Inc.: The Soovu Labs Inc. battery powered device is a one inch diameter heating pod that attaches to the user via a ring system. The device may be programmed to deliver a wide variety of treatment algorithms. Control of the devices are through a phone-based bluetooth connection. The treatment algorithm used for all subjects in this arm maintained a steady temperature of 37 degrees C.
Period: Overall Study
Arm/Group | High Level Pulsed Heat | Low Level Steady Heat
Started | 49 | 51
Completed | 49 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- High Level Pulsed Heat: Subjects randomized to this arm received a generation 5 device (Soovu Labs Inc.) that produced 30 minutes of heat. The heat was delivered as waves peaking at 45° C.
  Generation 5 device Soovu Labs Inc.: The Soovu Labs Inc. battery powered device is a one inch diameter heating pod that attaches to the user via a ring system. The device may be programmed to deliver a wide variety of treatment algorithms. Control of the devices are through a phone-based bluetooth connection.
- Low Level Steady Heat: Subjects randomized to this arm received an identical device (Soovu Labs Inc.) that produced 30 minutes ot heat. The heat was delivered in a steady manner at 37° C.
  Generation 5 device Soovu Labs Inc.: The Soovu Labs Inc. battery powered device is a one inch diameter heating pod that attaches to the user via a ring system. The device may be programmed to deliver a wide variety of treatment algorithms. Control of the devices are through a phone-based bluetooth connection.
- Total: Total of all reporting groups
Arm/Group | High Level Pulsed Heat | Low Level Steady Heat | Total
Number analyzed (Participants) | 49 | 51 | 100
Age, Categorical [Count of Participants; unit: Participants] — Starting Numerical Pain Score (NPS 0-10)
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 44 | 48 | 92
    >=65 years | 5 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 34 | 67
  Male | 16 | 17 | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 49 | 51 | 100
Numerical Pain Scale (NPS) [Mean (Standard Deviation); unit: units on a scale] — The Numeric Pain Scale is a 0-10 scale. It is validated over multiple populations and is a research standard for assessing pain.
  units on a scale | 5.56 (0.06) | 5.55 (0.07) | 5.55 (0.06)

OUTCOME MEASURES:

1. Primary Outcome: Pain Rating
Description: Numerical Pain Score (NPS) Range Zero (minimum) through ten (maximum score) thirty minutes after completion of the treatment session.
Time Frame: Changes in the Numerical Pain Scale will be compared between baseline and 30 minutes after minutes of treatment.
Measure: Mean (Standard Error); unit: reduction in pain score on a scale
Arm/Group | High Level Pulsed Heat | Low Level Steady Heat
Number analyzed (Participants) | 49 | 51
reduction in pain score on a scale | -1.40 (0.016) | -0.68 (0.019)
Statistical Analysis 1: Comparison: High Level Pulsed Heat vs Low Level Steady Heat; Demographic and clinical characteristics were tabulated by randomization group. The primary outcome was change in pain score from baseline to 30 minutes after treatment ended. Linear regression was used to compare differences in primary outcome between treatment and control groups adjusting for initial pain level. Unadjusted comparisons are also presented. Change in pain scores at each other post baseline time point were similarly analyzed; Test type: Other — The hypothesis is that the high level pulsed heat group will show statistically more pain relief than the low level steady heat group; p < 0.05, Regression, Linear; Linear regression was used to compare differences in primary outcome between treatment and control groups adjusting for initial pain level

2. Other Pre Specified Outcome: Pain Relief 30 Minutes After the Intervention
Description: Numerical Pain Scale Range Zero (minimum) through ten (maximum score) In this study a lower number on the Numeric Pain Scale means the subject(s) has less pain. Less pain particularly in the experimental group is a better outcome.
Time Frame: Changes in the Numerical Pain Scale will be compared between baseline and thirty minutes post intervention.
Population: All subjects with longstanding chronic low back pain median duration 10 years. Subjects who received the high level pulsed heat device with heat pulses up to 45 degrees C. Steady heat subjects received a device that heated to 37 degrees C at a steady level.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- High Level Pulsed Heat: Subjects who received the high level pulsed heat device with heat pulses up to 45 degrees C.
- Steady Heat Group: Subjects who received the steady heat device with heat received a steady level of heat at 37 degrees C.
Arm/Group | High Level Pulsed Heat | Steady Heat Group
Number analyzed (Participants) | 49 | 51
units on a scale | -1.40 (0.016) | -0.68 (0.019)

ADVERSE EVENTS:
Time Frame: 6 months including duration of study until mid November 2019
Groups:
- High Level Pulsed Heat: Subjects in this group received the active (experimental) device that utilized high level pulsed heat to a temperature of 45 degrees C.
- Low Level Steady Heat Group: Subjects in this group received the control device that utilized steady heat at a temperature of 37 degrees C.
Arm/Group | High Level Pulsed Heat | Low Level Steady Heat Group
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/51
Other Adverse Events (participants affected / at risk) | 0/49 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/03/NCT04109703/Prot_SAP_000.pdf